CLINICAL TRIAL: NCT03152487
Title: Randomized Trial Comparing Endoscopic Ultrasound-guided Radiofrequency Ablation vs.Endoscopic Ultrasound-guided Celiac Plexus Neurolysis in the Alleviation of Abdominal Pain in Patients With Pancreatic Cancer
Brief Title: Trial Comparing EUS-guided Radiofrequency Ablation vs. EUS-guided Celiac Plexus Neurolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1035541
Record Dates: First submitted 2017-04-20; First posted 2017-05-15 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Carcinoma Metastatic; Pancreatic Adenocarcinoma; Pancreatic Neoplasms; Pancreatic Cancer; Pancreatic Cancer, Adult
Keywords: endoscopic ultrasound; celiac plexus neurolysis; radiofrequency ablation; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic cancer, adult | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Subjects will randomized to either a group that receives Celiac Plexus Neurolysis or Radiofrequency Ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celiac Plexus Neurolysis (Active Comparator): CPN will be undertaken at the celiac space which is located between the aorta and the celiac artery origin. A 22 or 19-gauge Fine Needle Aspiration (FNA) needle is used, and its tip is placed slightly anterior and cephalic to the origin of the celiac artery. Aspiration is first performed using a syringe to ensure that vascular puncture has not occurred. 10 mL Bupivacaine is injected first, followed by 20 mL of 98% alcohol.
  Interventions: Other: Celiac Plexus Neurolysis
- Radiofrequency Ablation (Active Comparator): Once the celiac ganglia are identified on EUS, a 19-gauge FNA needle is inserted into the center of the ganglion or area of celiac plexus under EUS guidance. The radiofrequency (RF) probe (EMcision, Montreal, Canada) is advanced through the FNA needle. Radiofrequency ablation is performed via the probe for 90 seconds, followed by a 90 second rest and repeated as required.
  Interventions: Other: Radiofrequency Ablation

INTERVENTIONS:
Other: Celiac Plexus Neurolysis — This intervention involves accessing the Celiac Plexus Nerve via endoscopic guided ultrasound and then injecting the nerve bundle with bupivacaine.
  Arms: Celiac Plexus Neurolysis
Other: Radiofrequency Ablation — Radiofrequency ablation is performed via the probe for 90 seconds, followed by a 90 second rest. This is repeated until the entire ganglion becomes hyperechoic on EUS.
  Arms: Radiofrequency Ablation

SUMMARY:
Pancreatic cancer is the second most common gastrointestinal malignancy. Abdominal discomfort is a main symptom in patients with pancreatic cancer. Approximately 75% have pain at diagnosis and over 90% in advanced stages. Pain control is an important part of the plan of care for patients with pancreatic cancer.. The celiac plexus is a group of nerves that supply organs in the abdomen. EUS-guided celiac plexus neurolysis (EUS-CPN) has been widely used for pain management in patients with pancreatic cancer. Radiofrequency ablation of celiac ganglia or celiac plexus (EUS-RFA) is also being performed to alleviate abdominal pain in pancreatic cancer patients. However currently no comparative studies exist comparing EUS-CPN with EUS-RFA. The purpose of the study is to compare EUS-CPN with EUS-RFA for pain management in pancreatic patients, in order to determine which technique is better at improving pain in pancreatic cancer patients.

DETAILED DESCRIPTION:
Pancreatic cancer is the second most common gastrointestinal malignancy and fourth leading cause of cancer mortality. The incidence in the US is estimated at 8.8 per 100,000 population with 30,000 new cases diagnosed annually. The prognosis of unresectable pancreatic cancer is poor; overall 1 and 5-year survivals do not exceed 20 and 4%, respectively. For the minority of patients (15%) who are resectable at diagnosis, the median survival is 10-20 months, with 5-year survival of 10-25%.

Abdominal discomfort is a predominant symptom in patients with pancreatic cancer. Approximately 75% have pain at diagnosis and over 90% in advanced stages. Therefore a major aspect of palliation is provision of adequate pain control. The standard approach to pain management is based on the World Health Organization (WHO) 3-step ladder, beginning with non-opioid analgesics (e.g. non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen), followed by weak opioids and then finally strong opioids as necessary. Virtually all patients require escalating doses of opioids during their disease. Adjuvant therapies, including other medications (e.g. trazodone, tricyclic anti-depressants, and bisphosphonates), palliative radionucleotides, external beam radiation, or chemotherapy may also be useful for symptomatic control.

In the last 10 years, EUS-guided celiac plexus neurolysis (EUS-CPN) has been widely practiced for alleviation of pain in patients with pancreatic cancer and has been shown to be effective. At our institution, radiofrequency ablation (EUS-RFA), which involves ablation of celiac ganglia or celiac plexus using a radiofrequency catheter, is being performed to alleviate abdominal pain in pancreatic cancer patients. However currently no comparative studies exist comparing EUS-CPN with EUS-RFA for pain alleviation in pancreatic cancer patients.

In this randomized trial, the investigators will be comparing EUS-CPN with EUS-RFA for pain alleviation in pancreatic patients, in order to determine which technique is better at improving pain in pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. The subject is capable of understanding and complying with protocol requirements.
3. The subject is able to understand and willing to sign an informed consent form prior to the initiation of any study procedures.
4. Abdominal pain typical for pancreatic cancer
5. Cross-sectional imaging findings consistent with pancreatic cancer
6. Pancreatic cancer confirmed by EUS-FNA in patients referred for suspected pancreatic cancer OR Patients with known diagnosis of pancreatic cancer
7. Inoperable pancreatic cancer as determined during EUS or prior CT

Exclusion Criteria:

1. Age <19 years
2. Unable to obtain consent for the procedure from the patient
3. Unable to safely undergo EUS for any reason
4. Irreversible coagulopathy (Prothrombin time > 18 secs, platelet count < 50,000/ml)
5. Previous CPN or other neurolytic block that could affect pancreatic cancer-related pain or had implanted epidural or intrathecal analgesic therapy
6. Another cause for abdominal pain such as pseudocyst, ulcer or other intraabdominal disorder
7. Pregnant women will be excluded. This will be confirmed by self-report. Pregnancy in females of childbearing potential will be determined by routine preoperative urine or serum Human Chorionic Gonadotropin (HCG) testing.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Subject assessment of abdominal pain | Baseline to 4 week follow up
  Abdominal pain will be assessed with pain scores from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Pancreatic Cancer module (QLQ-PAN26). The questionnaire has 26 questions with scoring ranging from a minimum of 26 to a maximum of 104. The higher the score, the worse the subject's quality of life rating.

SECONDARY OUTCOMES:
Subject assessment of Quality of Life. | Baseline; 2 week follow up; 4 week follow up
  Quality of life (QOL) as assessed by the quality of life instrument: the Functional Assessment of Cancer Therapy, Pancreatic Cancer (FACT-PA) (i.e. QLQ-30 and PAN-26)
Narcotic Use | Initial visit; 2 week follow up; 4 week follow up
  Subjects will be asked about their medication usage to manage pain and the answers will be documented.
Crossover to alternate technique | 48 hours post procedure; 2 week follow up; 4 week follow up
  Cross-over to the alternate technique due to inadequate response to the original technique (defined as < 50% decrease in VAS score post-original technique).
Adverse effects, and endoscopic adverse events | 48 hours post procedure; 2 week follow up; 4 week follow up
  Information regarding complications if any, that the subject may have experienced, which can include hypotension, diarrhea, neuropathic pain, paraplegia and endoscopic adverse events
Survival rate | 2 week follow up; 4 week follow up
  Information regarding if the subject is alive or deceased.
Pain per the VAS tool. | Baseline; 48 hour post procedure; 2 week follow up; 4 week follow up
  Abdominal pain will be assessed with a standardized 11-point continous visual analog pain scale (with "0" equaling no pain, "5" moderate pain and "10" worst pain ever.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam S Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD).

REFERENCES:
- [Background] Yan BM, Myers RP. Neurolytic celiac plexus block for pain control in unresectable pancreatic cancer. Am J Gastroenterol. 2007 Feb;102(2):430-8. doi: 10.1111/j.1572-0241.2006.00967.x. Epub 2006 Nov 13. PMID 17100960
- [Background] Carr DB, Goudas LC, Balk EM, Bloch R, Ioannidis JP, Lau J. Evidence report on the treatment of pain in cancer patients. J Natl Cancer Inst Monogr. 2004;(32):23-31. doi: 10.1093/jncimonographs/lgh012. PMID 15263038
- [Background] World Health Organization. Cancer pain relief, 2nd Ed. Geneva: WHO, 2006
- [Background] Penman ID, Rosch T; EUS 2008 Working Group. EUS 2008 Working Group document: evaluation of EUS-guided celiac plexus neurolysis/block (with video). Gastrointest Endosc. 2009 Feb;69(2 Suppl):S28-31. doi: 10.1016/j.gie.2008.11.004. No abstract available. PMID 19179165
- [Background] Gunaratnam NT, Sarma AV, Norton ID, Wiersema MJ. A prospective study of EUS-guided celiac plexus neurolysis for pancreatic cancer pain. Gastrointest Endosc. 2001 Sep;54(3):316-24. doi: 10.1067/mge.2001.117515. PMID 11522971
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Kastler A, Aubry S, Sailley N, Michalakis D, Siliman G, Gory G, Lajoie JL, Kastler B. CT-guided stellate ganglion blockade vs. radiofrequency neurolysis in the management of refractory type I complex regional pain syndrome of the upper limb. Eur Radiol. 2013 May;23(5):1316-22. doi: 10.1007/s00330-012-2704-y. Epub 2012 Nov 9. PMID 23138389
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Bang JY, Hasan MK, Sutton B, Holt BA, Navaneethan U, Hawes R, Varadarajulu S. Intraprocedural increase in heart rate during EUS-guided celiac plexus neurolysis: Clinically relevant or just a physiologic change? Gastrointest Endosc. 2016 Nov;84(5):773-779.e3. doi: 10.1016/j.gie.2016.03.1496. Epub 2016 Apr 2. PMID 27048974
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Derived] Bang JY, Sutton B, Hawes RH, Varadarajulu S. EUS-guided celiac ganglion radiofrequency ablation versus celiac plexus neurolysis for palliation of pain in pancreatic cancer: a randomized controlled trial (with videos). Gastrointest Endosc. 2019 Jan;89(1):58-66.e3. doi: 10.1016/j.gie.2018.08.005. Epub 2018 Aug 16. PMID 30120957